CLINICAL TRIAL: NCT05432947
Title: A Pilot Comparison of 68Ga-P16-093 and 18F-FDG PET/CT Imaging in the Same Group of Clear Cell Renal Cell Carcinoma Patients
Brief Title: 68Ga-P16-093 and 18F-FDG PET/CT Imaging in the Same Group of Clear Cell Renal Cell Carcinoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH NM-RCC
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-09

CONDITIONS: Clear Cell Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-P16-093 and 18F-FDG PET/ CT scan (Experimental): Within 1 week, each patient underwent PET/CT scan after intravenous administration of 68Ga-P16-093 and 18F-FDG, respectively.
  Interventions: Drug: 68Ga-P16-093; Drug: 18F-FDG

INTERVENTIONS:
Drug: 68Ga-P16-093 — Intravenous injection of 68Ga-P16-093 with a dosage of 1.8-2.2 MBq (0.05-0.06 mCi)/kg.
  Other Names: 68Ga-P16-093 injection
Drug: 18F-FDG — Intravenous injection of 18F-FDG with a dosage of 5.55 MBq (0.15 mCi)/kg.
  Other Names: 18F-FDG injection

SUMMARY:
PSMA is highly expressed on the cell surface of the microvasculature of several solid tumors, including clear cell renal cell carcinoma (ccRCC). This makes it a potentially imaging target for the detection of ccRCC. This pilot study was designed to evaluate the diagnostic performance of 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, which was compared with 18F-FDG PET/CT in the same group of ccRCC patients.

DETAILED DESCRIPTION:
Renal cell carcinoma (RCC) is the most common solid tumor within the kidney and accounts for approximately 3% of all malignancies in the world. Clear cell RCC (ccRCC) is the most common subtype and accounts for the majority of kidney cancer-related deaths. Importantly, pro-angiogenic factors (VEGF, PDGF) are strongly upregulated in clear cell RCC, leading to high vascularized tumors. Prostate-specific membrane antigen (PSMA), as known as folate hydrolase I or glutamate carboxypeptidase II, is overexpressed on the cells of prostatic adenocarcinoma. However, PSMA is also expressed by tumor cells or neovascular endothelial cells of various solid neoplasms, such as renal cell carcinoma. Therefore, PSMA may be an ideal target for the diagnosis of ccRCC. 68Ga-P16-093, a novel radiopharmaceutical targeting PSMA, with the urea fragment of a conjugate that employs the HBED-CC chelator for labeling with 68Ga(III). The HBED-based chelating ligand binds the 68Ga3+ ion with high affinity in a pseudo-octahedral N2O4 coordination sphere by its two phenolate O, two amino-acetate carboxylate O, and two amino N donor atoms. This pilot study was designed to evaluate the diagnostic performance of 68Ga-P16-093 in the same group of ccRCC patients, compared with 18F-FDG PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* patients with confirmed or suspected clear cell Renal cell carcinoma;
* 68Ga-P16-093 18F-FDG PET/CT within a week;
* signed written consent.

Exclusion Criteria:

* pregnancy;
* breastfeeding;
* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance | through study completion, an average of 1 year
  comparing the number of tumor detected by 68Ga-P16-093 and 18F-FDG PET/CT

SECONDARY OUTCOMES:
standardized uptake value (SUV) of tumor | through study completion, an average of 1 year
  comparing the SUVmax of tumor derived from 68Ga-P16-093 and 18F-FDG PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang G, Li L, Wang J, Zang J, Chen J, Xiao Y, Fan X, Zhu L, Kung HF, Zhu Z. Head-to-head comparison of [68Ga]Ga-P16-093 and 2-[18F]FDG PET/CT in patients with clear cell renal cell carcinoma: a pilot study. Eur J Nucl Med Mol Imaging. 2023 Apr;50(5):1499-1509. doi: 10.1007/s00259-022-06101-3. Epub 2023 Jan 5. PMID 36600099